CLINICAL TRIAL: NCT06543368
Title: Low-Cost Platelet-Rich Plasma Injection for the Management of Hemarthropathy
Brief Title: Low-Cost Platelet-Rich Plasma for Hemarthropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Daniel Cushman, Principal Investigator, Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00177846
Record Dates: First submitted 2024-07-29; First posted 2024-08-09 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Hemarthrosis; Hemophilia
Keywords: Hemophilia; Hemarthrosis; PRP; Platelet Rich Plasma
MeSH Terms: conditions — Hemarthrosis; Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRP Injection (Experimental): 45mL of blood is drawn from the subject in a standard-of-care manner into 3 x 20mL syringes, each containing 2mL of sodium citrate (anticoagulant). Each syringe is prepared and capped, then placed into a centrifuge. The resulting separated blood is then drawn off into a single new sterile syringe, which can be used for the injection. Blood and PRP analysis: We will perform a full analysis (a complete blood count [CBC] with differential) on subjects' whole blood and their prepared LC-PRP. Importantly, we will include all data required in the PRP minimum reporting standards, including "platelet, differential leukocyte, and red cell analysis of all samples."
  Interventions: Biological: Intra articular PRP Injection

INTERVENTIONS:
Biological: Intra articular PRP Injection — A total of 20 joints (estimated 10-15 patients) will receive injections, performed at day 0 and 3 weeks, for a total of two injections - two injections have demonstrated superior outcomes to one, and will increase our number of injections to improve the proof of feasibility. All subjects will receive ultrasound-guided intra-articular joint injections by an experienced sports medicine provider after local anesthesia with 1% lidocaine to the extra-articular structures, namely the skin and joint capsule, to increase comfort.

SUMMARY:
Orthopedic complications can be injuries or diseases that affect the bones, muscles, and joints. Hemarthropathy is due to bleeding disorders, most commonly hemophilia, and can result in severe issues related to chronic amounts of blood in the body's joints. This causes swelling, pain, and loss of joint function. A serious barrier to treating many patients with bleeding disorders creates higher health risks and costs. Platelet-rich plasma (PRP) injection is a method that can reduce the cost of care while still offering a similar standard of care for patients.

This study intends to show that low-cost PRP can be done safely in patients with bleeding disorders, without the need for expensive equipment, while monitoring patient treatment results. Study participants will receive injections for joint conditions. Being in the study requires attending 1 to 2 in-person visits at the study clinic. Participants will also complete surveys using email, text messages, in person, and/or on the phone. Participation lasts about 6 months.

DETAILED DESCRIPTION:
This study will be performed as a prospective, single arm study. Consecutive patients eligible for a standard-of-care injection will be enrolled from the Utah Center for Bleeding and Clotting Disorders. The University of Utah non-operative sports medicine team currently performs hundreds of injections monthly, and the PI works closely with the orthopedic complaints of patients with bleeding disorders. From a research standpoint, the investigators have successfully performed numerous randomized controlled prospective trials on a variety of musculoskeletal conditions in the past and have already validated this method on a large cohort of patients with knee osteoarthritis (OA).

Potential subjects will then be approached by a member of the research team to discuss the consideration of taking part in the study if they meet the inclusion criteria of this study project. Using all forms of good clinical practice, a member of the study team will review with the participant the Informed Consent Form, allow participant to read the informed consent (ICF) and ask questions prior to signing the ICF. Potential subjects may also be asked by other physicians or staff members familiar with the study.

Low Cost-Platelet Rich Plasma (LC-PRP) preparation method: See Documents for full details. This method follows the same procedures as the standard-of-care, FDA-cleared method used by numerous commercial machines; thus it does not require additional FDA clearance or approval. To summarize the full method in the appendix, 45mL of blood is drawn from the subject in a standard-of-care manner into 3 x 20mL syringes, each containing 2mL of sodium citrate (anticoagulant). Each syringe is prepared and capped, then placed into a centrifuge. The resulting separated blood is then drawn off into a single new sterile syringe, which can be used for the injection. Blood and PRP analysis: The investigators will perform a full analysis (a complete blood count (CBC) with differential) on subjects' whole blood and their prepared LC-PRP. Importantly, the investigators will include all data required in the PRP minimum reporting standards, including "platelet, differential leukocyte, and red cell analysis of all samples." Also note that although the investigators are collecting these values for the purposes of the study, CBC values are not needed in the community.

Injections: A total of 20 joints (estimated 10-15 patients) will receive injections, performed at day 0 and 3 weeks, for a total of two injections - two injections have demonstrated superior outcomes to one, and will increase our number of injections to improve the proof of feasibility. All subjects will receive ultrasound-guided intra-articular joint injections by an experienced sports medicine provider after local anesthesia with 1% lidocaine to the extra-articular structures, namely the skin and joint capsule, to increase comfort. Note: though the investigators are using ultrasound guidance to ensure that they are guaranteeing accurate injectate placement for this study, this is not necessarily required in the community setting. These will be performed after the patient's typical factor infusions, if applicable.

Questionnaire: The investigators will collect demographic information along with baseline and subsequent functional patient reported outcomes, namely the WOMAC (knee), FAOS (ankle), and the QuickDASH (elbow). REDCap will be used to administer surveys and store data. The investigators will additionally ask about adverse events, pain, global satisfaction, global injection satisfaction, and medications.

Data collection time points and follow-up: Follow-up data (see timeline below) will be administered electronically. Subjects will be queried by email, text message, in person, and/or by telephone regarding treatment outcomes at 0, 1, 3, and 6 months after the second injection. Three months will be the primary endpoint, and six months will be an exploratory, unfunded endpoint.

* LC-PRP Outcomes: As this is a feasibility study, it is likely that this study will be underpowered for clinical outcomes. However, the investigators will still monitor pain and the above outcome measures and identify potential time-related improvements.
* Economic Evaluation: The investigators will track staff-, time-, equipment-, and supply-related costs to accurately identify costs associated with each injection. This will ensure that costs are accurately recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any adult age with symptomatic hemarthropathy of the ankle, knee, or elbow, based on radiographs within the last 24 months.
* Patients must have failed at least six weeks of conventional conservative treatments (such as medication or physical therapy).

Exclusion Criteria:

* Exclusion criteria will include recent (last two years) surgery to the affected joint, prior joint replacement.
* Prior orthobiologic injection into the affected joint.
* Thrombocytopenia
* Inability to receive factor prior to PRP injection.
* Active systemic or local infection at the site of injection,
* Non-ambulatory patients
* Body mass index (BMI) over 50
* Recent (six month) or current corticosteroid injection/intake.

Patients with hemarthropathy in multiple joints will be eligible for up to 2 joints if multiple fit the criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-07-23 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Pain (numeric pain rating system) | 6-months
  Prospectively evaluate clinical outcomes in a cohort of patients with bleeding disorders for pain over six months (at baseline, 1, 3, and 6 months), numeric pain rating system (0-10).

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 6-months
  WOMAC at baseline, 1, 3, and 6 months for participants receiving knee injections. The questionnaire consists of 24 questions, divided into these three categories (pain, stiffness, and physical function). Patients rate their symptoms on a scale from 0 (no pain or difficulty) to 4 (extreme pain or difficulty).
Quick Disabilities of Arm Shoulder and Hand (QuickDASH) | 6-months
  QuickDASH at baseline, 1, 3, and 6 months for participants receiving elbow injections. The QuickDASH consists of 11 questions, each with five response options ranging from "no difficulty" to "unable". You rate your symptoms and functional abilities based on the past week. A higher score indicates greater disability.
Foot and Ankle Outcome Score (FAOS) | 6-months
  FAOS at baseline, 1, 3, and 6 months for participants receiving ankle injections. The FAOS is a questionnaire with 42 questions, each rated on a 5-point Likert scale (0-4). Higher scores indicate better function and less pain. The total score ranges from 0 to 100, with higher scores representing better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Nie LY, Zhao K, Ruan J, Xue J. Effectiveness of Platelet-Rich Plasma in the Treatment of Knee Osteoarthritis: A Meta-analysis of Randomized Controlled Clinical Trials. Orthop J Sports Med. 2021 Mar 2;9(3):2325967120973284. doi: 10.1177/2325967120973284. eCollection 2021 Mar. PMID 33718505
- [Background] Chu J, Duan W, Yu Z, Tao T, Xu J, Ma Q, Zhao L, Guo JJ. Intra-articular injections of platelet-rich plasma decrease pain and improve functional outcomes than sham saline in patients with knee osteoarthritis. Knee Surg Sports Traumatol Arthrosc. 2022 Dec;30(12):4063-4071. doi: 10.1007/s00167-022-06887-7. Epub 2022 Feb 6. PMID 35124707
- [Background] Dai WL, Zhou AG, Zhang H, Zhang J. Efficacy of Platelet-Rich Plasma in the Treatment of Knee Osteoarthritis: A Meta-analysis of Randomized Controlled Trials. Arthroscopy. 2017 Mar;33(3):659-670.e1. doi: 10.1016/j.arthro.2016.09.024. Epub 2016 Dec 22. PMID 28012636
- [Background] Tan J, Chen H, Zhao L, Huang W. Platelet-Rich Plasma Versus Hyaluronic Acid in the Treatment of Knee Osteoarthritis: A Meta-analysis of 26 Randomized Controlled Trials. Arthroscopy. 2021 Jan;37(1):309-325. doi: 10.1016/j.arthro.2020.07.011. Epub 2020 Jul 15. PMID 32679294
- [Background] Baria MR, Vasileff WK, Borchers J, DiBartola A, Flanigan DC, Plunkett E, Magnussen RA. Treating Knee Osteoarthritis With Platelet-Rich Plasma and Hyaluronic Acid Combination Therapy: A Systematic Review. Am J Sports Med. 2022 Jan;50(1):273-281. doi: 10.1177/0363546521998010. Epub 2021 Apr 8. PMID 33831332
- [Background] Gualtierotti R, Solimeno LP, Peyvandi F; Ultrasound in hemophilic arthropathy study group. Ultrasound evaluation of hemophilic arthropathy: a proposal of definitions in a changing landscape. Res Pract Thromb Haemost. 2024 Jan 3;8(1):102314. doi: 10.1016/j.rpth.2023.102314. eCollection 2024 Jan. PMID 38322151
- [Background] Caviglia H, Landro ME, Daffunchio C, Galatro G, Douglas Price AL, Salgado P, Neme D. Platelet Rich Plasma for Chronic Synovitis Treatment in Patients with Haemophilia. Haemophilia. 2017 Jul;23(4):613-619. doi: 10.1111/hae.13212. Epub 2017 May 4. PMID 28470911
- [Background] Piuzzi NS, Ng M, Kantor A, Ng K, Kha S, Mont MA, Muschler GF. What Is the Price and Claimed Efficacy of Platelet-Rich Plasma Injections for the Treatment of Knee Osteoarthritis in the United States? J Knee Surg. 2019 Sep;32(9):879-885. doi: 10.1055/s-0038-1669953. Epub 2018 Sep 6. PMID 30189436
- [Background] Chu CR, Rodeo S, Bhutani N, Goodrich LR, Huard J, Irrgang J, LaPrade RF, Lattermann C, Lu Y, Mandelbaum B, Mao J, McIntyre L, Mishra A, Muschler GF, Piuzzi NS, Potter H, Spindler K, Tokish JM, Tuan R, Zaslav K, Maloney W. Optimizing Clinical Use of Biologics in Orthopaedic Surgery: Consensus Recommendations From the 2018 AAOS/NIH U-13 Conference. J Am Acad Orthop Surg. 2019 Jan 15;27(2):e50-e63. doi: 10.5435/JAAOS-D-18-00305. PMID 30300216
- [Background] D'Angiolella LS, Cortesi PA, Rocino A, Coppola A, Hassan HJ, Giampaolo A, Solimeno LP, Lafranconi A, Micale M, Mangano S, Crotti G, Pagliarin F, Cesana G, Mantovani LG. The socioeconomic burden of patients affected by hemophilia with inhibitors. Eur J Haematol. 2018 Oct;101(4):435-456. doi: 10.1111/ejh.13108. Epub 2018 Jul 27. PMID 29889317
- [Background] O'Hara J, Hughes D, Camp C, Burke T, Carroll L, Diego DG. The cost of severe haemophilia in Europe: the CHESS study. Orphanet J Rare Dis. 2017 May 31;12(1):106. doi: 10.1186/s13023-017-0660-y. PMID 28569181
- [Background] Beitzel K, Allen D, Apostolakos J, Russell RP, McCarthy MB, Gallo GJ, Cote MP, Mazzocca AD. US definitions, current use, and FDA stance on use of platelet-rich plasma in sports medicine. J Knee Surg. 2015 Feb;28(1):29-34. doi: 10.1055/s-0034-1390030. Epub 2014 Sep 30. PMID 25268794
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] McAlindon TE, Bannuru RR, Sullivan MC, Arden NK, Berenbaum F, Bierma-Zeinstra SM, Hawker GA, Henrotin Y, Hunter DJ, Kawaguchi H, Kwoh K, Lohmander S, Rannou F, Roos EM, Underwood M. OARSI guidelines for the non-surgical management of knee osteoarthritis. Osteoarthritis Cartilage. 2014 Mar;22(3):363-88. doi: 10.1016/j.joca.2014.01.003. Epub 2014 Jan 24. PMID 24462672
- [Background] Singh H, Knapik DM, Polce EM, Eikani CK, Bjornstad AH, Gursoy S, Perry AK, Westrick JC, Yanke AB, Verma NN, Cole BJ, Chahla JA. Relative Efficacy of Intra-articular Injections in the Treatment of Knee Osteoarthritis: A Systematic Review and Network Meta-analysis. Am J Sports Med. 2022 Sep;50(11):3140-3148. doi: 10.1177/03635465211029659. Epub 2021 Aug 17. PMID 34403285
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Tavassoli M, Janmohammadi N, Hosseini A, Khafri S, Esmaeilnejad-Ganji SM. Single- and double-dose of platelet-rich plasma versus hyaluronic acid for treatment of knee osteoarthritis: A randomized controlled trial. World J Orthop. 2019 Sep 18;10(9):310-326. doi: 10.5312/wjo.v10.i9.310. eCollection 2019 Sep 18. PMID 31572668
- [Background] Chen CX, Baker JR, Nichol MB. Economic Burden of Illness among Persons with Hemophilia B from HUGS Vb: Examining the Association of Severity and Treatment Regimens with Costs and Annual Bleed Rates. Value Health. 2017 Sep;20(8):1074-1082. doi: 10.1016/j.jval.2017.04.017. Epub 2017 Jun 17. PMID 28964439
- [Background] Saxena K. Barriers and perceived limitations to early treatment of hemophilia. J Blood Med. 2013 May 16;4:49-56. doi: 10.2147/JBM.S43734. Print 2013. PMID 23700376
- [Background] Laver L, Marom N, Dnyanesh L, Mei-Dan O, Espregueira-Mendes J, Gobbi A. PRP for Degenerative Cartilage Disease: A Systematic Review of Clinical Studies. Cartilage. 2017 Oct;8(4):341-364. doi: 10.1177/1947603516670709. Epub 2016 Sep 1. PMID 28317389
- [Background] Patel S, Gahlaut S, Thami T, Chouhan DK, Jain A, Dhillon MS. Comparison of Conventional Dose Versus Superdose Platelet-Rich Plasma for Knee Osteoarthritis: A Prospective, Triple-Blind, Randomized Clinical Trial. Orthop J Sports Med. 2024 Feb 26;12(2):23259671241227863. doi: 10.1177/23259671241227863. eCollection 2024 Feb. PMID 38410168
- [Background] Poenaru D, Sandulescu MI, Cinteza D. Intraarticular management of chronic haemophilic arthropathy (Review). Biomed Rep. 2023 Jul 21;19(3):59. doi: 10.3892/br.2023.1641. eCollection 2023 Sep. PMID 37614987
- [Background] Rodriguez-Merchan EC. Intra-articular injection of platelet-rich plasma in patients with hemophilia and painful knee joint cartilage degeneration. Expert Rev Hematol. 2023 Jun;16(6):407-416. doi: 10.1080/17474086.2023.2166922. Epub 2023 Jan 12. PMID 36609192
- [Background] Teyssler P, Kolostova K, Bobek V. The impact of platelet-rich plasma on chronic synovitis in hemophilia. Acta Orthop Belg. 2014 Mar;80(1):11-7. PMID 24873079
- [Background] Li TY, Wu YT, Chen LC, Cheng SN, Pan RY, Chen YC. An exploratory comparison of single intra-articular injection of platelet-rich plasma vs hyaluronic acid in treatment of haemophilic arthropathy of the knee. Haemophilia. 2019 May;25(3):484-492. doi: 10.1111/hae.13711. Epub 2019 Mar 13. PMID 30866117
- [Background] Gualtierotti R, Solimeno LP, Peyvandi F. Hemophilic arthropathy: Current knowledge and future perspectives. J Thromb Haemost. 2021 Sep;19(9):2112-2121. doi: 10.1111/jth.15444. Epub 2021 Jul 27. PMID 34197690
- [Background] Cuesta-Barriuso R, Donoso-Ubeda E, Merono-Gallut J, Ucero-Lozano R, Perez-Llanes R. Hemophilic Arthropathy: Barriers to Early Diagnosis and Management. J Blood Med. 2022 Oct 17;13:589-601. doi: 10.2147/JBM.S343924. eCollection 2022. PMID 36277171
- [Background] van Vulpen LFD, Thomas S, Keny SA, Mohanty SS. Synovitis and synovectomy in haemophilia. Haemophilia. 2021 Feb;27 Suppl 3(Suppl 3):96-102. doi: 10.1111/hae.14025. Epub 2020 Jun 3. PMID 32490595
- [Background] Elksnins-Finogejevs A, Vidal L, Peredistijs A. Intra-articular platelet-rich plasma vs corticosteroids in the treatment of moderate knee osteoarthritis: a single-center prospective randomized controlled study with a 1-year follow up. J Orthop Surg Res. 2020 Jul 10;15(1):257. doi: 10.1186/s13018-020-01753-z. PMID 32650801
- [Background] Forogh B, Mianehsaz E, Shoaee S, Ahadi T, Raissi GR, Sajadi S. Effect of single injection of platelet-rich plasma in comparison with corticosteroid on knee osteoarthritis: a double-blind randomized clinical trial. J Sports Med Phys Fitness. 2016 Jul-Aug;56(7-8):901-8. Epub 2015 Jul 14. PMID 26173792
- [Background] Joshi Jubert N, Rodriguez L, Reverte-Vinaixa MM, Navarro A. Platelet-Rich Plasma Injections for Advanced Knee Osteoarthritis: A Prospective, Randomized, Double-Blinded Clinical Trial. Orthop J Sports Med. 2017 Feb 13;5(2):2325967116689386. doi: 10.1177/2325967116689386. eCollection 2017 Feb. PMID 28255569
- [Background] Habib GS. Systemic effects of intra-articular corticosteroids. Clin Rheumatol. 2009 Jul;28(7):749-56. doi: 10.1007/s10067-009-1135-x. Epub 2009 Feb 28. PMID 19252817
- [Background] Belk JW, Kraeutler MJ, Houck DA, Goodrich JA, Dragoo JL, McCarty EC. Platelet-Rich Plasma Versus Hyaluronic Acid for Knee Osteoarthritis: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Am J Sports Med. 2021 Jan;49(1):249-260. doi: 10.1177/0363546520909397. Epub 2020 Apr 17. PMID 32302218
- [Background] Laudy AB, Bakker EW, Rekers M, Moen MH. Efficacy of platelet-rich plasma injections in osteoarthritis of the knee: a systematic review and meta-analysis. Br J Sports Med. 2015 May;49(10):657-72. doi: 10.1136/bjsports-2014-094036. Epub 2014 Nov 21. PMID 25416198
- [Background] O'Dowd A. Update on the Use of Platelet-Rich Plasma Injections in the Management of Musculoskeletal Injuries: A Systematic Review of Studies From 2014 to 2021. Orthop J Sports Med. 2022 Dec 9;10(12):23259671221140888. doi: 10.1177/23259671221140888. eCollection 2022 Dec. PMID 36532150
- [Background] Xiong Y, Gong C, Peng X, Liu X, Su X, Tao X, Li Y, Wen Y, Li W. Efficacy and safety of platelet-rich plasma injections for the treatment of osteoarthritis: a systematic review and meta-analysis of randomized controlled trials. Front Med (Lausanne). 2023 Jun 27;10:1204144. doi: 10.3389/fmed.2023.1204144. eCollection 2023. PMID 37441691